CLINICAL TRIAL: NCT00465829
Title: Longitudinal Assessment of Bariatric Surgery (LABS-2)
Brief Title: Long-term Effects of Bariatric Surgery
Acronym: LABS-2
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven Belle, Professor, University of Pittsburgh
Other Study IDs: DK6657_2; U01DK066557 (NIH)
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of LABS-2 is to use standardized techniques and measures to assess the longer-term safety and efficacy of bariatric surgery by:

1. comparing post-surgical outcomes to pre-operative status
2. examining risks and benefits of surgery.

LABS-2 will determine the associations between clinical/demographic patient characteristics, components of the surgical procedure, and peri-operative and post-operative care with post-operative risks and changes in patient status.

Funds are not available to pay for the surgery for patients, only to address research questions.

DETAILED DESCRIPTION:
The primary goal of LABS-2 is to evaluate the efficacy and safety of bariatric surgery over a longer term than LABS-1, i.e., more than 30 days. Using a sample of the LABS-1 cohort, approximately 2,400 patients, will be recruited over 3 years. LABS-2 will include clinical assessments and detailed interviews and questionnaires pre-operatively and at several post-operative time points (30 days, 6 months, 12 months following surgery, and annually thereafter) to assess risks of surgery, and changes in clinical, metabolic, and psychosocial characteristics in patients, and health care utilization following bariatric surgery. Detailed data about the surgical procedure and peri- and post-operative care will also be collected to determine if components of the surgical procedure, and peri-operative and post-operative care as well as clinical/demographic patient characteristics are associated with post-operative risks and changes in patient status. Patients enrolled in LABS-2 will provide blood specimens pre-operatively and post-operatively to address LABS-2 hypotheses and additional samples will be stored at the NIDDK tissue repository for serologic, pathologic and genomic testing of other hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age and undergo bariatric surgery by a LABS certified surgeon
* Previous enrollment in LABS-1
* Selected by algorithm to be included in LABS-2

Exclusion Criteria:

* Informed consent not obtained
* Prior bariatric surgery
* Unlikely to comply with follow-up protocol
* Unable to communicate with local study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All bariatric surgical candidates at participating LABS centers who are 18 years or older and have not had prior bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2458 (Actual)
Dates: Start 2006-03; Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Berk, MD, Principal Investigator — Columbia University; Anita Courcoulas, MD,MPH,FACS, Principal Investigator — University of Pittsburgh Medical Center; David R Flum, MD,MPH,FACS, Principal Investigator — University of Washington; James E Mitchell, MD, Principal Investigator — Neuropsychiatric Research Institute; Bruce M Wolfe, MD,FACS, Principal Investigator — Oregon Health and Science University; Walter J Pories, MD,FACS, Principal Investigator — East Carolina Medical Center
Locations (9):
- United States (9):
  - Cornell University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Neuropsychiatric Research Institute, Fargo, North Dakota
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data deposited in NIDDK funded data repository

REFERENCES:
- [Derived] White GE, Courcoulas AP, Broskey NT, Rogan SC, Jeyabalan A, King WC. Maternal and Neonatal Outcomes of Pregnancy within 7 years after Roux-Y Gastric Bypass or Sleeve Gastrectomy Surgery. Obes Surg. 2023 Jun;33(6):1764-1772. doi: 10.1007/s11695-023-06575-6. Epub 2023 Apr 4. PMID 37014543
- [Derived] Wolfe MB, Williams TJ, Dewey EN, Mitchell JE, Pomp A, Wolfe BM. Health change awareness and its association with weight loss following bariatric surgery. Health Psychol. 2023 Jun;42(6):403-410. doi: 10.1037/hea0001279. Epub 2023 Mar 27. PMID 36972088
- [Derived] Purnell JQ, Dewey EN, Laferrere B, Selzer F, Flum DR, Mitchell JE, Pomp A, Pories WJ, Inge T, Courcoulas A, Wolfe BM. Diabetes Remission Status During Seven-year Follow-up of the Longitudinal Assessment of Bariatric Surgery Study. J Clin Endocrinol Metab. 2021 Mar 8;106(3):774-788. doi: 10.1210/clinem/dgaa849. PMID 33270130
- [Derived] Smith KE, Mason TB, Cao L, Crosby RD, Steffen KJ, Garcia L, King WC, Mitchell JE. Trajectories of depressive symptoms and relationships with weight loss in the seven years after bariatric surgery. Obes Res Clin Pract. 2020 Sep-Oct;14(5):456-461. doi: 10.1016/j.orcp.2020.08.007. Epub 2020 Sep 12. PMID 32933863
- [Derived] Bjornstad P, Nehus E, Jenkins T, Mitsnefes M, Moxey-Mims M, Dixon JB, Inge TH. Five-year kidney outcomes of bariatric surgery differ in severely obese adolescents and adults with and without type 2 diabetes. Kidney Int. 2020 May;97(5):995-1005. doi: 10.1016/j.kint.2020.01.016. Epub 2020 Feb 3. PMID 32229096
- [Derived] Dewberry LC, Jalivand A, Gupta R, Jenkins TM, Beamish A, Inge TH, Courcoulas A, Helmrath M, Brandt ML, Harmon CM, Chen M, Dixon JB, Zeller M, Michalsky MP. Weight Loss and Health Status 5 Years After Adjustable Gastric Banding in Adolescents. Obes Surg. 2020 Jun;30(6):2388-2394. doi: 10.1007/s11695-020-04504-5. PMID 32124210
- [Derived] Heshka S, Lemos T, Astbury NM, Widen E, Davidson L, Goodpaster BH, DeLany JP, Strain GW, Pomp A, Courcoulas AP, Lin S, Janumala I, Yu W, Kang P, Thornton JC, Gallagher D. Resting Energy Expenditure and Organ-Tissue Body Composition 5 Years After Bariatric Surgery. Obes Surg. 2020 Feb;30(2):587-594. doi: 10.1007/s11695-019-04217-4. PMID 31617114
- [Derived] Steffen KJ, King WC, White GE, Subak LL, Mitchell JE, Courcoulas AP, Flum DR, Strain G, Sarwer DB, Kolotkin RL, Pories W, Huang AJ. Changes in Sexual Functioning in Women and Men in the 5 Years After Bariatric Surgery. JAMA Surg. 2019 Jun 1;154(6):487-498. doi: 10.1001/jamasurg.2018.1162. PMID 30785625
- [Derived] Davidson LE, Yu W, Goodpaster BH, DeLany JP, Widen E, Lemos T, Strain GW, Pomp A, Courcoulas AP, Lin S, Janumala I, Thornton JC, Gallagher D. Fat-Free Mass and Skeletal Muscle Mass Five Years After Bariatric Surgery. Obesity (Silver Spring). 2018 Jul;26(7):1130-1136. doi: 10.1002/oby.22190. Epub 2018 May 30. PMID 29845744
- [Derived] Courcoulas AP, King WC, Belle SH, Berk P, Flum DR, Garcia L, Gourash W, Horlick M, Mitchell JE, Pomp A, Pories WJ, Purnell JQ, Singh A, Spaniolas K, Thirlby R, Wolfe BM, Yanovski SZ. Seven-Year Weight Trajectories and Health Outcomes in the Longitudinal Assessment of Bariatric Surgery (LABS) Study. JAMA Surg. 2018 May 1;153(5):427-434. doi: 10.1001/jamasurg.2017.5025. PMID 29214306
- [Derived] Menke MN, King WC, White GE, Gosman GG, Courcoulas AP, Dakin GF, Flum DR, Orcutt MJ, Pomp A, Pories WJ, Purnell JQ, Steffen KJ, Wolfe BM, Yanovski SZ. Contraception and Conception After Bariatric Surgery. Obstet Gynecol. 2017 Nov;130(5):979-987. doi: 10.1097/AOG.0000000000002323. PMID 29016506
- [Derived] King WC, Chen JY, Belle SH, Courcoulas AP, Dakin GF, Elder KA, Flum DR, Hinojosa MW, Mitchell JE, Pories WJ, Wolfe BM, Yanovski SZ. Change in Pain and Physical Function Following Bariatric Surgery for Severe Obesity. JAMA. 2016 Apr 5;315(13):1362-71. doi: 10.1001/jama.2016.3010. PMID 27046364
- [Derived] Courcoulas AP, Christian NJ, O'Rourke RW, Dakin G, Patchen Dellinger E, Flum DR, Melissa Kalarchian PD, Mitchell JE, Patterson E, Pomp A, Pories WJ, Spaniolas K, Steffen K, Wolfe BM, Belle SH. Preoperative factors and 3-year weight change in the Longitudinal Assessment of Bariatric Surgery (LABS) consortium. Surg Obes Relat Dis. 2015 Sep-Oct;11(5):1109-18. doi: 10.1016/j.soard.2015.01.011. Epub 2015 Jan 23. PMID 25824474
- [Derived] Mitchell JE, King WC, Chen JY, Devlin MJ, Flum D, Garcia L, Inabet W, Pender JR, Kalarchian MA, Khandelwal S, Marcus MD, Schrope B, Strain G, Wolfe B, Yanovski S. Course of depressive symptoms and treatment in the longitudinal assessment of bariatric surgery (LABS-2) study. Obesity (Silver Spring). 2014 Aug;22(8):1799-806. doi: 10.1002/oby.20738. Epub 2014 Mar 25. PMID 24634371
- [Derived] Courcoulas AP, Christian NJ, Belle SH, Berk PD, Flum DR, Garcia L, Horlick M, Kalarchian MA, King WC, Mitchell JE, Patterson EJ, Pender JR, Pomp A, Pories WJ, Thirlby RC, Yanovski SZ, Wolfe BM; Longitudinal Assessment of Bariatric Surgery (LABS) Consortium. Weight change and health outcomes at 3 years after bariatric surgery among individuals with severe obesity. JAMA. 2013 Dec 11;310(22):2416-25. doi: 10.1001/jama.2013.280928. PMID 24189773
- [Derived] Mackey RH, Belle SH, Courcoulas AP, Dakin GF, Deveney CW, Flum DR, Garcia L, King WC, Kuller LH, Mitchell JE, Pomp A, Pories WJ, Wolfe BM; Longitudinal Assessment of Bariatric Surgery Consortium Writing Group. Distribution of 10-year and lifetime predicted risk for cardiovascular disease prior to surgery in the longitudinal assessment of bariatric surgery-2 study. Am J Cardiol. 2012 Oct 15;110(8):1130-7. doi: 10.1016/j.amjcard.2012.05.054. Epub 2012 Jun 27. PMID 22742719
- See also: Study web site — http://www.niddklabs.org